CLINICAL TRIAL: NCT04074070
Title: Prevalence of Sonographic Abnormalities of Joints and Entheses in Patients With Psoriasis With or Without Musculoskeletal Complains
Brief Title: Prevalence of Sonographic Abnormalities of Joints and Entheses in Psoriasis Patients With or Without Musculoskeletal Complains
Acronym: EchoPso
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190683; 2018-A02781-54 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-08-19; First posted 2019-08-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis
Keywords: psoriasis; psoriatic arthritis; ultrasound
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriasis with and without musculoskeletal complains: psoriasis with and without musculoskeletal complains
  Interventions: Other: Ultrasound examination
- Healthy individuals
  Interventions: Other: Ultrasound examination
- Psoriatic arthritis
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Ultrasound examination of joints, tendons and entheses.

SUMMARY:
The objectives of this study are:

* to estimate the prevalence and severity of inflammatory (synovitis, tenosynovitis, enthesitis, dactylitis) and structural (erosions, osteophytes, enthesophytes, cortical irregularities ) ultrasound lesions in psoriasis patients with or without related musculoskeletal symptoms;
* to compare them to healthy subjects or patients suffering from rheumatoid arthritis and osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Psoriasis diagnosed by a dermatologist;
* Able to participate in the study;
* Informed consent signed.

Exclusion Criteria:

- Chronic disease likely to cause musculoskeletal symptoms (connective tissue diseases, inflammatory bowel diseases, overload disorders, crystal related arthritis, septic arthritis...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients consulting the dermatology department of Ambroise Paré hospital for cutaneous psoriasis between September 2019 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
synovitis | through study completion, an average of 1 year
  Number and percentage, N (%) of patients with at least one synovitis.
enthesitis | through study completion, an average of 1 year
  N (%) of patients with at least one ultrasound enthesitis.
joint erosion | through study completion, an average of 1 year
  N (%) of patients with at least one joint erosion.
osteophyte/ cortical irregularity | through study completion, an average of 1 year
  N (%) of patients with at least one osteophyte/ cortical irregularity.
enthesophyte | through study completion, an average of 1 year
  N (%) of patients with at least one enthesophyte.

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Antonietta D'Agostino, MD, PhD, Principal Investigator — Rheumatology Department, Ambroise Paré Hospital
Locations (1):
- Rheumatology Department, Ambroise Paré Hospital, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No